CLINICAL TRIAL: NCT03144388
Title: Task-specificity for Locomotor Recovery Following SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, George Hornby, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU1705279110
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Parallel-group with optional crossover
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors at each measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable Stepping Training (Experimental): High intensity stepping training in multiple environments, including overground, on a treadmill and on stairs.
  Interventions: Procedure: Variable Stepping Training
- Variable Non-specific Training (Active Comparator): High intensity non-stepping training, including balance, strength, and cycling tasks
  Interventions: Procedure: Variable Non-specific Training

INTERVENTIONS:
Procedure: Variable Stepping Training — Six weeks (20 sessions) of high intensity stepping training in multiple variable environments
  Arms: Variable Stepping Training
Procedure: Variable Non-specific Training — Six weeks (20 sessions) of high intensity stepping training in multiple variable environments
  Arms: Variable Non-specific Training

SUMMARY:
The primary goal of the proposed study is to identify the contributions of the amount of task-specific practice on locomotor (i.e., walking) recovery in patients with chronic (> 1 yr) motor incomplete spinal cord injury (iSCI). Consistent with principles of motor learning and exercise physiology, the investigators contend that certain training (i.e., dosage) parameters of physical rehabilitation are critical to mobility outcomes following neurological injury. Specifically, the specificity, amount and intensity of physical interventions (i.e., practice) may influence specific outcomes in the patient population treated. In ambulatory patients with iSCI, there are very few studies that have controlled for or targeted these training variables or their influence on locomotor recovery. Previous work suggests these training parameters may influence locomotor recovery in patients with other neurological disorders (i.e., stroke), although few studies have attempted to delineate similar contributions of in iSCI. Indeed, no studies have carefully controlled the amount of task-specific practice during physical rehabilitation of patients with iSCI, and such interventions are rarely utilized in the clinical setting. The goal of the present study is to delineate the relative contributions of amount of task-specific training on locomotor outcomes in individuals with iSCI. Using a cross-over, randomized clinical trial design, the investigators anticipated non-specific (i.e., non-stepping) training activities would result in smaller improvements as compared to task-specific (stepping) training. The investigators will investigate the effects of such training on walking performance and kinematics, as well as the impairments thought to contribute to walking performance. Successful completion of this project could have an immediate impact on rehabilitation research and treatment of people following iSCI, and may be utilized to treat more subacute patients with iSCI or other acute-onset neurological disorders.

DETAILED DESCRIPTION:
The primary goal of the proposed study is to identify the contributions of the amount of task-specific practice on locomotor (i.e., walking) recovery in patients with chronic (> 1 yr) motor incomplete spinal cord injury (iSCI). The investigators will do this by building on previous work directed towards identifying the essential exercise training parameters that maximize locomotor recovery. Consistent with principles of motor learning and exercise physiology, the investigators contend that certain training (i.e., dosage) parameters of physical rehabilitation, including the type (specificity) and amount of task practice, are critical to mobility outcomes following neurological injury. Previous work suggests these training parameters may influence locomotor recovery in patients with other neurological disorders (i.e., stroke), although few studies have attempted to delineate similar contributions of amount of task-specific practice in iSCI. Indeed, no studies have carefully controlled these training parameters during physical rehabilitation of patients with iSCI, and such interventions are rarely utilized in the clinical setting.

Reasons for these knowledge gaps from other rehabilitation studies to patients with iSCI or lack of clinical implementation are unclear, but may be due to adherence to traditional rehabilitation theories. One concern is that practicing only stepping tasks reduces attention towards hallmark physical impairments following iSCI, such as loss of strength or postural stability, which are considered primary determinants of decreased mobility. Only a few studies have addressed whether providing only structured stepping training can mitigate these impairments without their explicit practice, but not in the iSCI population. A related concern is that focused stepping training without significant attention towards impairments or gait quality may exaggerate altered movement strategies, which could be reinforced with repeated practice. However, there is little data to suggest "worsening" of abnormal gait patterns following high intensity training. Rather, recent findings suggest patients demonstrate more normal kinematics. If focused task specific (i.e., stepping) training is to be applied clinically, the investigators must delineate its contributions towards improving locomotor function, and their effects on underlying impairments and gait kinematics.

The central hypotheses are that stepping training in iSCI results in:1) greater locomotor gains as compared to non-specific interventions; 2) gains in selected impairments underlying gait dysfunction (i.e., strength and metabolic capacity and efficiency); and, 3) improvements in gait quality. To test these hypotheses, the proposed crossover, assessor-blinded, randomized clinical trial (RCT) is designed to test the effects of specificity of rehabilitation training applied early-post-stroke. In this RCT, patients > 1 year post-iSCI will be allocated to 4-6 weeks (20 session) of high-intensity stepping training or high-intensity non-specific training. Importantly, training intensity will be held constant to account for this potential confounding factor. Blinded assessments will be performed prior to and following each training paradigm. The investigators will address 3 specific aims:

Specific Aim 1: Demonstrate that high intensity stepping training in patients with chronic iSCI produces greater locomotor gains as compared to high intensity non-specific training strategies.

Hypothesis 1: High intensity stepping training will result in greater increases in gait speeds and distances Specific Aim 2: Test the effects of these training strategies on impairments and non-locomotor mobility tasks.

Hypothesis 2: Higher intensity stepping training groups will result in greater gains in metabolic capacity and efficiency.

Specific Aim 3: Analyze the potential effects of high intensity stepping or non-specific training on gait quality.

Hypothesis 3: High intensity training will result in improved sagittal-plane gait kinematics consistent with normal locomotor function, due in part to greater locomotor speeds, as compared to non-specific training strategies.

The aims represent an innovative approach to improving long-term mobility outcomes of patients with iSCI by applying selected principles of motor learning and exercise physiology yet untested in this population. Expected outcomes will be demonstration of the efficacy of a high intensity stepping training paradigm, with further understanding of potential underlying mechanisms and movement strategies used with improved locomotor performance. Successful completion of this project could have an immediate impact on rehabilitation research and treatment of people following iSCI, and may be utilized to treat more subacute patients with iSCI

ELIGIBILITY:
Inclusion Criteria:

* individuals with chronic (>1 yr duration) motor iSCI at the level or T10 (anatomical) or above
* ages 18-75 years
* ability to walk without physical assistance but with below-knee braces and assistive devices as needed
* self-selected gait speeds between 0.01-1.0 m/s.
* not currently receiving physical therapy

Exclusion Criteria:

* uncontrolled cardiopulmonary or metabolic disease that limits exercise participation
* active heterotopic ossification
* recurrent history of lower extremity fractures
* previous orthopedic or other peripheral or central neurological injury that may impair locomotor function
* history of botulinum toxin injection < 3 months prior
* Patients who are prescribed intrathecal or oral anti-spastics should agree to limit changes in anti-spastic use throughout the training and testing period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Walking Speed | change in walking speed from baseline testing to post-testing following 6 weeks of training
  fastest comfortable walking speed over short distances

SECONDARY OUTCOMES:
Walking Distance | change in walking speed from baseline testing to post-testing following 6 weeks of training
  distance covered over 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hornby, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Data available as requested